CLINICAL TRIAL: NCT06446843
Title: Assessment of Injectable Platelet-rich Fibrin With Hyaluronic Acid Versus Hyaluronic Acid in Management of Temporomandibular Joint Internal Derangement
Brief Title: Platelet-Rich Fibrin and Hyaluronic Acid vs. Hyaluronic Acid Injection for TMJ Internal Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Baghdad Mohammed abdo-alhage, Principal researcher at oral and Maxillofacial surgery department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethical approval no.: 12 4 24
Record Dates: First submitted 2024-06-02; First posted 2024-06-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Internal Derangement
Keywords: Hyaluronic acid; Injectable PRF; TMJ Internal derangement; Temporomandibular joint

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (control group) (Active Comparator): arthrocentesis with Ringer's lactate solution, of the superior joint compartment
  Interventions: Combination Product: (Arthrocentesis followed by i-PRF +HA)
- (study group1) (Experimental): arthrocentesis with Ringer's lactate solution, of the superior joint compartment then inject 1ml of HA.
  Interventions: Combination Product: (Arthrocentesis followed by i-PRF +HA)
- (study group2) (Experimental): arthrocentesis with Ringer's lactate solution, of the superior joint compartment then inject
  1 ml of i- PRF then1ml of HA following arthrocentesis.
  Interventions: Combination Product: (Arthrocentesis followed by i-PRF +HA)

INTERVENTIONS:
Combination Product: (Arthrocentesis followed by i-PRF +HA) — Intra-articular I-PRF with HA will be injected in the joint,1 ml of I-PRF will be injected inside the joint, Then from 25mg/ml of HA , 1ml will be injected into the superior joint space

SUMMARY:
Injectable PRF technology, according to literature evidence, ensures the release of growth factors over time which play a major role in the release of regenerative factors for tissue repair after injection, while HA is an anti-inflammatory medication that can provide rapid relief from pain and inflammation in joints. It is a major natural component of synovial fluid that plays an important role in lubrication of synovial tissues However, its effect is typically temporary, and it doesn't promote tissue healing or regeneration.

For this reason, this protocol has been designed with the aim to investigate whether injection in the injection i- pRF with HA can achieve the same improvements of pain and function, compare this technique with arthrocentesis.

DETAILED DESCRIPTION:
One group will receive arthrocentesis only, the second group will receive 1 mm hyaluronic acid injection and the third group will receive a mixture of 1 ml hyaluronic acid, 1 ml of injectable PRF

ELIGIBILITY:
Inclusion Criteria:

* Presence of TMJ-ID related symptoms.
* Patients suffering from TMJ internal derangement (disc displacement with reduction).
* Age limit between 20 and 45years so Patient less than 21years will need assent form …as well as written informed consent from the parents \guardians.
* No previous TMJ surgical procedures
* Acquisition of informed consent.
* Cooperative patient
* Patients free from any systemic disease that may affect the procedure.

Exclusion Criteria:

* Previous malignant head and neck neoplasms.
* Patients suffering from inflammatory or connective tissue systemic diseases.
* Neurologic disorders.
* History of bony or fibrous adhesion
* Gross mechanical restrictions and condylar fractures, previous TMJ surgery, TMJ ankylosis, or acute infection.
* Patients maintained on anti-coagulants, muscle relaxants, non-steroidal anti-inflammatory drugs within 48 h preoperatively, corticosteroid injection at treatment site within one month or systemic use of corticosteroids within 2 weeks was also excluded in this study.
* Uncooperative patient
* Pregnant and lactating female.
* Patients with systemic diseases (e.g., rheumatoid arthritis, psoriatic arthritis, or juvenile arthritis), and those who had shown symptoms of hypersensitivity to the HA solution.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
pain intensity at TMJ during spontaneous mouth opening and with articular palpation and forced opening | evaluated at the preoperative examination (baseline) and reassessed at follow-up evaluation at 1 month, 3, month, and 6 months after the procedure.
  Pain measured through a (10 scale) visual analogue scale (VAS)
Maximum mouth opening | evaluated at the preoperative examination (baseline) and reassessed at follow-up evaluation at 1 month, 3, month, and 6 months after the procedure.
  mandibular mouth opening defined as MIO (maximum interincisal opening) >/35

SECONDARY OUTCOMES:
MRI disc angle changes | preoperative examination (baseline) and 6 months after the procedure.
  MRI unit :degree of angle between the posterior margin of the disc and the vertical line drawn through the Centre of the condyle.

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Kadry, Study Director — Associate professor at Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

REFERENCES:
- [Background] Yuce E, Komerik N. Comparison of the Efficiacy of Intra-Articular Injection of Liquid Platelet-Rich Fibrin and Hyaluronic Acid After in Conjunction With Arthrocentesis for the Treatment of Internal Temporomandibular Joint Derangements. J Craniofac Surg. 2020 Oct;31(7):1870-1874. doi: 10.1097/SCS.0000000000006545. PMID 32433129
- [Background] Ghoneim NI, Mansour NA, Elmaghraby SA, Abdelsameaa SE. Treatment of temporomandibular joint disc displacement using arthrocentesis combined with injectable platelet rich fibrin versus arthrocentesis alone. J Dent Sci. 2022 Jan;17(1):468-475. doi: 10.1016/j.jds.2021.07.027. Epub 2021 Aug 21. PMID 35028072
- [Background] Harba AN, Harfoush M. Evaluation of the participation of hyaluronic acid with platelet-rich plasma in the treatment of temporomandibular joint disorders. Dent Med Probl. 2021 Jan-Mar;58(1):81-88. doi: 10.17219/dmp/127446. PMID 33847473
- [Background] Hegab AF, Hameed HIAA, Hassaneen AM, Hyder A. Synergistic effect of platelet rich plasma with hyaluronic acid injection following arthrocentesis to reduce pain and improve function in TMJ osteoarthritis. J Stomatol Oral Maxillofac Surg. 2023 Feb;124(1S):101340. doi: 10.1016/j.jormas.2022.11.016. Epub 2022 Nov 19. PMID 36414172
- [Background] Isik G, Kenc S, Ozveri Koyuncu B, Gunbay S, Gunbay T. Does the Use of Injectable Platelet-Rich Fibrin After Arthrocentesis for Disc Displacement Without Reduction Improve Clinical Outcomes? J Oral Maxillofac Surg. 2023 Jun;81(6):689-697. doi: 10.1016/j.joms.2023.02.014. Epub 2023 Mar 13. PMID 36924792
- [Background] Toameh MH, Alkhouri I, Karman MA. Management of patients with disk displacement without reduction of the temporomandibular joint by arthrocentesis alone, plus hyaluronic acid or plus platelet-rich plasma. Dent Med Probl. 2019 Jul-Sep;56(3):265-272. doi: 10.17219/dmp/109329. PMID 31577070